CLINICAL TRIAL: NCT01702467
Title: A Single-Blind, Randomized, Placebo-Controlled Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single, Oral Escalating Doses of GSK2647544 in Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single, Oral Escalating Doses of GSK2647544 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 116698
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Alzheimer's Disease
Keywords: Lp-PLA2; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease | interventions — GSK2647544

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSK2647544 (Experimental): The starting dose of GSK2647544 is 0.5 mg. The escalating doses to be administered will be determined based on study results from previous dose (s).
  Interventions: Drug: GSK2647544
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK2647544 — Capsules containing 0.5mg to 50mg of GSK2647544.
  Arms: GSK2647544
Drug: Placebo — Matching placebo capsules.
  Arms: Placebo

SUMMARY:
The current study will examine the safety, tolerability, plasma pharmacokinetics (PK), and plasma pharmacodynamics (PD) of single-doses of GSK2647544.The study will be conducted as a randomized, single-blind, placebo controlled, 4-way crossover single oral ascending dose design in 2 independent cohorts, eight healthy male subjects in each of the cohorts. Each potential subject will undergo Screening visit, Treatment Phase and Follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males who are 18 to 55 years of age, inclusive
* Healthy as determined by a responsible and experienced physician
* aspartate aminotransferase (AST), Alanine transaminase (ALT), alkaline phosphatase and bilirubin <= 1.5xUpper Limit of Normal (ULN)
* Average of triplicate QTcB values and average of triplicate QTcF values must both < 450 millisecond (msec)
* Body weight > 50 kg (110 pounds) and body mass index (BMI) between 19 and 30
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods
* Capable of giving written informed consent

Exclusion Criteria:

* Those with Lp-PLA2 activity <=20 nanomole/minute/milliliter (mL)(for subjects with 2 known birth parents of at least 50% Japanese, Chinese, or Korean ancestry)
* History of asthma, anaphylaxis or anaphalactoid reactions, severe allergic responses
* History of hypercoagulable state or history of thrombosis
* A history of biliary tract disease including a history of liver disease with elevated liver function tests of known or unknown etiology
* Positive Human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C at screening
* History of regular use of tobacco- or nicotine-containing products within three months of the study and/or has a positive breath CO at screening
* History of alcohol consumption exceeding, on average, 21 drinks/week for men (1 drink = 100 mL of wine or 240 mL of beer or 30 mL of hard liquor in Australia) within 6 months of the first dose of study medication
* Positive urine drug or positive breath alcohol test at screening or at admission to Clinical Research Unit
* Unable to refrain from use of prescription or non-prescription drugs and vitamins within 7 days or 5 half-lives (whichever is longer) prior to administration of study
* Unable to refrain from use of dietary/herbal supplements including (but not limited to) St. John's wort, kava, ephedra (ma huang), gingko biloba, DHEA, yohimbe, saw palmetto, ginseng and red yeast rice within 14 days prior to treatment with study medication
* Treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) prior to dosing
* Unable to refrain from consumption of grapefruit or grapefruit juice within 7 days prior to the first dose of study medication
* For male subjects, an unwillingness to abstain from sexual intercourse with pregnant or lactating women or an unwillingness to use a condom plus partner use of a highly effective contraceptive if engaging in sexual intercourse with a woman who could become pregnant until discharge from the study
* Donation of blood in excess of 500 mL within 56 days prior to dosing
* History of sensitivity to heparin or heparin-induced thrombocytopenia
* Subjects, who in the investigator's judgement, pose a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behaviour and/or any suicidal ideation of type 4 or 5 on the C-SSRS in the last 6 months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-10-19 (Actual); Primary Completion 2013-05-15 (Actual); Study Completion 2013-05-15 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GSK2647544 as assessed by number of subjects with adverse events (AE)s | 5 days in each of the 4 dosing session
  Safety and tolerability parameters will include recording of AEs
Safety and tolerability of GSK2647544 as assessed by change from Baseline in laboratory values | 5 days in each of the 4 dosing session
  Safety and tolerability parameters will include laboratory (haematology, clinical chemistry, urinalysis) values at Screening, Day -1, Day 3 and Follow-up (7-14 days post-last dose)
Safety and tolerability of GSK2647544 as assessed by change from Baseline in ECG readings | 5 days in each of the 4 dosing session
  Safety and tolerability parameter will include the electrocardiogram (ECG) readings at Screening, Day -1, Day 1, Day 2, Day 3 and Follow-up (7-14 days post-last dose)
Safety and tolerability of GSK2647544 as assessed by change from Baseline in Telemetry ECG parameters | 3 Days in each of the 4 dosing session
  Safety and tolerability parameter will include the Telemetry ECG readings from 30 minutes pre-dosing till 48 hours post-dosing
Safety and tolerability of GSK2647544 as assessed by change from Baseline in vital signs | 5 days in each of the 4 dosing session
  Vital signs measurement include systolic and diastolic blood pressure and pulse rate at Screening, Day -1, Day 1, Day 2, Day 3, Day 4 and Follow-up (7-14 days post-last dose)
Safety and tolerability of GSK2647544 as assessed by using the Columbia Suicide Severity Rating Scale (C-SSRS) | 5 days in each of the 4 dosing session
  C-SSRS will be measured at Screening, Day -1, Day 1 (conducted prior to discharge) and Follow-up (7-14 days post-last dose)

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) of GSK2647544 | 4 Days in each of the 4 dosing session
  To assess PK profile of GSK2647544, Cmax of GSK2647544 will be measured
Time of peak plasma concentration (tmax) of GSK2647544 | 4 Days in each of the 4 dosing session
  To assess PK profile of GSK2647544 tmax of GSK2647544 will be measured
Area under the time concentration curve (AUC) of GSK2647544 | 4 Days in each of the 4 dosing session
  To assess PK profile of GSK2647544 AUC of GSK2647544 will be measured
Terminal half-life (t½ ) of GSK2647544 | 4 Days in each of the 4 dosing session
  To assess PK profile of GSK2647544 t½ of GSK2647544 will be measured
Apparent oral clearance (CL/F) of GSK2647544 | 4 Days in each of the 4 dosing session
  To assess PK profile of GSK2647544 CL/F of GSK2647544 will be measured
Predose plasma lipoprotein-associated phospholipase A2 (Lp-PLA2) activity and postdose Lp-PLA2 activity | 5 Days in each of the 4 dosing session
  It will be measured at Day 1, Day 2, Day 3, Day 4 and Day 5

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 116698 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116698?search=study&search_terms=116698#rs
- Available data/document: Clinical Study Report: 116698 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116698 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116698 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116698 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116698 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116698 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116698 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register